CLINICAL TRIAL: NCT07255196
Title: Virtual Vs Telephone Education in Radiotherapy - Randomized Clinical Trial
Brief Title: Virtual Vs Telephone Education in Radiotherapy
Acronym: VIPER-RT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Michael Velec, Clinician Scientist - Radiation Therapist, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-5883
Record Dates: First submitted 2025-11-17; First posted 2025-11-28 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Patient Education; Radiotherapy
Keywords: Virutal Care; Videoconferencing; Patient Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care Arm (No Intervention): 30 minute radiation therapist-led pre-treatment education with a telephone call to explain upcoming radiotherapy treatment, side-effects, appointment logistics and answer patient questions
- Videoconferencing Arm (Active Comparator): 45 minute radiation therapist-led pre-treatment education with a videoconferencing call to explain upcoming radiotherapy treatment, side-effects, appointment logistics and answer patient questions
  Interventions: Device: Videoconferencing Software for Pre-Treatment Education

INTERVENTIONS:
Device: Videoconferencing Software for Pre-Treatment Education — Videoconferencing software used for pre-treatment education with face-to-face, patient-to-provider communication using a slide deck with images to help with pre-treatment educational material for radiotherapy
  Arms: Videoconferencing Arm

SUMMARY:
The goal of this clinical trial is to compare whether the use of videoconferencing in breast cancer patients undergoing radiotherapy is better for pre-treatment education than telephone calls. The main question it aims to answer is in breast cancer patient receiving radiotherapy, does videoconferencing, compared to telephone calls for pre-treatment education result in decreased procedural fears and concerns? The investigators hypothesize that the use of videoconferencing for pre-treatment radiotherapy education will decrease breast cancer patients' procedural fears and concerns. Researchers will compare the current standard of care in a 30 minute radiation therapist led pre-treatment education call to the intervention of a 45 minute radiation therapist led videoconferencing call to see if the intervention reduces patient procedural fears and concerns, anxiety levels, and has higher patient satisfaction. Participants will be asked to complete questionnaires at three time points: 1. Baseline - at time of study consent. 2. CT-Simulation - after their radiotherapy CT-Simulation appointment. 3. Day 1 Treatment - after their first day of radiotherapy treatment.

DETAILED DESCRIPTION:
Rationale: Breast cancer (BC) is a major health concern worldwide. In 2024, it was stated that breast cancer makes up almost 25% of all new cancer diagnoses in women. Breast cancer was also found to be the leading cause of cancer death in women. The use of Radiation Therapy (RT) plays a major role in the treatment of breast cancer. Although RT has such a large role, the complexity of RT can be psychologically and physically demanding for patients. Many patients require and seek out a large amount of information to help facilitate understanding of RT. Evidence suggests the use of a pre-treatment education session led by a Radiation Therapist(s) has been found to reduce patients' procedural fears, concerns and overall anxiety levels. Since the COVID-19 pandemic, telephone calls became the standard for pre-treatment education. Recently a study by Magliozzi et al has found the use of videoconferencing-based education demonstrated higher levels of patient satisfaction and preference over telephone. However, evidence directly comparing these two modalities against each other is lacking.

Objective: The aim of this study is comparing the effectiveness of the current standard in pre-RT education using telephone calls versus videoconferencing led education in reducing breast cancer patients' procedural fears and concerns related to RT. The investigators hypothesize that the use of videoconferencing will decrease breast cancer patients' procedural concerns more than using telephone calls. If videoconferencing does reduce breast cancer patients' procedural fears and concerns, future directions for radiation therapy education will be to implement videoconferencing as the current standard for breast cancer patients, and eventually all patients. In addition to this, cancer centers worldwide will be able to implement a virtual approach if the cancer center has the resources to do such.

Experimental Approach: To test this hypothesis, the experimental approach is a prospective randomized clinical trial of Radiation Therapist-led patient education sessions comparing the two modalities, videoconferencing and telephone. Breast cancer patients receiving radical breast radiotherapy above the age of 18 and have a device with access to the internet and Microsoft Teams will be consented and randomized 1:1 into the intervention group (videoconferencing) or control group (telephone). The primary endpoint for this study is a change in patients' procedural fears and concerns using the Cancer Treatment Survey (CaTS). A total sample size of 130 patients, measured at 3 time points (T1: baseline, T2: post CT-Simulation, and T3: post day 1 treatment), will achieve 80% power at a 0.05 significance level to detect a mean difference of 0.44 in the CaTS procedural fears and concerns subscale between groups using a repeated measures design. Secondary endpoints for this study include patient reported anxiety levels measured by the Hospital Anxiety and Depression Scale, anxiety subscale (HADS-A), and overall patient satisfaction measured using a survey adapted from Berlin et al. Anxiety levels will be measured at all three time points, whereas satisfaction will be measured at T2 due to its close timing with the education session.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Access to an internet connected device with a microphone and camera
* Able to communicate in English with/without a translator
* Receiving radical breast cancer radiotherapy

Exclusion Criteria:

* Previous radiotherapy treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Cancer Treatment Survey Procedural Fears & Concerns Subscale (CaTS-PC) | Measured at three time points (T1-T3). T1: Baseline, T2: exactly after patient CT-Simulation and T3: exactly after patient first day of radiotherapy
  11 total questions relating to patients procedural fears and concerns on a Likert-scale (1-5), mean scores are taken from this to generate a procedural fear and concern level out of 5, with lower scores indicating less procedural fears and concerns

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS-A) | Measured at three time points (T1-T3). T1: Baseline, T2: exactly after patient CT-Simulation and T3: exactly after patient first day of radiotherapy
  7 question survey measured on a 4 point scale (0-3). Total scores are summed and give a indication of patient anxiety levels at the time of completion based. Scores are divided as follows: 0-7 is considered normal, 8-10 is borderline or mild anxiety, and 11-21 is considered severe.
Satisfaction with Pre-Treatment Radiation Therapy Education Survey | Delivered at T2 - exactly after CT-Simulation
  6 likert scale question survey looking at patients overall satisfaction with the specific modality used for pre-treatment education. Looking at the overall appointment, as well as the informational needs of patients. Each question will be looked at individually.

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Center, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-07-21): https://cdn.clinicaltrials.gov/large-docs/96/NCT07255196/Prot_000.pdf